CLINICAL TRIAL: NCT06031350
Title: Peripapillary and Macular Vascular Changes of Unilateral Anterior Ischemic Optic Neuropathy: An Optical Coherence Tomography Angiography Study
Status: Completed | Type: Observational
Sponsor: Omar Said (Other)
Responsible Party: Sponsor-Investigator, Omar Said, Assistant professor of Ophthalmology, Fayoum University
Organization: Fayoum University (Other)
Other Study IDs: EOM64
Record Dates: First submitted 2023-09-02; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Non-arteritic Ischemic Optic Neuropathy
Keywords: OCTA AION NAION

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Diseased eyes: The 30 diseased eyes of the patients were considered the case group.
  Interventions: Diagnostic Test: Optical Coherence Tomography Angiography
- Fellow eyes: The 30 fellow eyes of the patients were considered the control group.
  Interventions: Diagnostic Test: Optical Coherence Tomography Angiography

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography Angiography — Optovue, Inc., Fremont, CA, USA

SUMMARY:
This series aims at studying the peripapillary and macular vascular changes in subjects with unilateral anterior ischemic optic neuropathy via Optical Coherence Tomography Angiography (OCTA).

DETAILED DESCRIPTION:
After approval of the local institutional ethics committee and local institutional review board, This study was conducted upon 30 patients diagnosed with acute NAION attending at Ophthalmology outpatient clinic in Fayoum University Hospitals. The participants were informed about the objectives of the study, the examination, investigations and the confidentiality of their information and their right not to participate in the study. OCT and OCTA was done for all subjects and control group with Optovue, Inc., Fremont, CA, USA. Patients were examined on presentation, after 6 weeks and lastly after 3 months. OCT was used for evaluation of Central macular thickness (CMT), nerve fiber layer thickness (NFLT) and ganglion cell complex (GCC). OCTA was done for quantitative evaluation of vessel density in the following: optic nerve head and peripapillary area, macular superficial vessel density, macular deep vessel density and foveal avascular zone. Vessel density was reported as the percentage of the total area that was occupied by blood vessels. All parameters were calculated automatically by the machine software. Poor quality scans and those with motion artifacts were excluded. Statistical analysis was performed using SPSS software (version 22; SPSS, Chicago, IL, USA). The data were presented as the mean ± SD values. P-value <0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with unilateral NAION and acute or sudden painless drop of vision.
* A normal fellow eye.
* Age ≥ 40 years old.

Exclusion Criteria:

* Arteritic type of AION.
* NAION patients in chronic phase.
* Acute phase NAION patients with any other optic neuropathy in the other eye.
* Eyes with opaque media.
* Elevated intraocular pressure (>22 mmHg).
* Refractive errors greater than 6 diopters of spherical equivalent.
* Poor cooperation with fixation or the OCTA examination.

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients presenting to the outpatient clinic of the department of Ophthalmology in Fayoum university hospitals with unilateral acute NAION. 30 patients (60 eyes) divided into 2 groups: 30 NAION eyes as the case group, and 30 fellow eyes as a control group.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Peripapillary and macular vascular changes | 3 months (0,6,12 weeks)
  comparing vessel density in different areas and sectors of diseased and fellow eyes

SECONDARY OUTCOMES:
Thickness of different retinal layers | 3 months (0,6,12 weeks)
  comparing thickness of Central macular thickness (CMT), nerve fiber layer thickness (NFLT) and ganglion cell complex (GCC)

CONTACTS AND LOCATIONS:
Overall Officials: Omar Said, MD, Study Director — Assistant professor of Ophthalmology
Locations (1):
- Faculty of Medicine, Fayoum University, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided